CLINICAL TRIAL: NCT07310550
Title: Physical Therapy Program for Selective Motor Control
Brief Title: A Physical Therapy Program Targeting Lower Extremity Selective Motor Control in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Eileen Fowler, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0414
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Spastic Cerebral Palsy
Keywords: cerebral palsy; spastic; physical therapy; selective motor control; intervention; corticospinal tracts
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor for GMFM was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants who have the intervention (Experimental): physical therapy exercise intervention
  Interventions: Other: Selective movement of individual lower limb joints; Other: Knee joint strengthening at high velocities; Other: Ankle controlled gaming; Other: Functional activities based on child and parental goals; Other: Sensori-motor exercises

INTERVENTIONS:
Other: Selective movement of individual lower limb joints — Children practices moving the joints of each lower leg independently.
Other: Knee joint strengthening at high velocities — In sitting, the thigh and trunk are secured to a seat and the lower leg to a moving arm that provides resistance at exercise velocities progressing up to a maximum of 300 deg/s.
Other: Ankle controlled gaming — With the child in sitting, the ankle is secured to a moving segment. The child can control games such as tennis by dorsiflexing and plantar flexing their ankle at increasing velocities to meet the demands of the game.
Other: Functional activities based on child and parental goals — The Canadian Occupational Performance Measure is used to identify functional goals. Activities to address these goals are designed by physical therapists and practiced during camp.
Other: Sensori-motor exercises — Walking barefoot over sand and grass. Foot and ankle sensory exploration using materials with various textures.

SUMMARY:
The goal of this intervention study is to learn whether a physical therapy exercise camp called will improve leg movement (motor control) and functional ability in children with spastic CP who are between 5 and 18 years. The main questions the study aims to answer are:

* Does the ability to move the knee at high velocities improve?
* Does function such as walking, running, hopping, climbing stairs improve?
* Will the brain tracts that control movement change?
* Will children who have better independent control of joint motion improve more?

All participants will:

* Attend 15 sessions of an exercise camp for 3 hours per day
* Perform a home exercise program after the camp ends

Measurements:

* Lower extremity selective motor control
* Knee muscle strength at high speeds using an exercise machine
* Gross motor function
* Gait analysis (walking patterns)
* Parent's perception of their child's ability and their satisfaction with that ability
* Change in brain motor tracts using a scanner (MRI) for participants that meet the inclusion criteria for MRI

MRI measurements will be taken twice (before and immediately after the treatment). All other measurements and will be taken 3 times (before, immediately after the treatment and approximately 4 months after the treatment).

ELIGIBILITY:
Inclusion Criteria:

* spastic cerebral palsy
* age between 5-18 years
* ability to walk at least 10 meters
* ability to follow simple verbal directions

Exclusion Criteria:

All participants

* botulinum toxin or serial casting within the preceding 3 months
* recent orthopedic or neurological surgery within the preceding 12 months
* uncontrolled seizures

For participants undergoing MRI

* inability to lie still
* incompatible metal implants
* baclofen pumps or shunts

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure | nine months
  Children are asked to perform functional activities including standing, walking, running, balancing and stair climbing. The data are entered into a computer program to create a score ranging from 0-100. A higher score indicates better function.

SECONDARY OUTCOMES:
Knee joint torque | nine months
  Three repetitions of maximum effort knee extension and flexion torque are collected at 0-300 deg/s for the affected lower limbs. Outcomes are the percent of knee joints that can produce measurable torque at each velocity and the peak joint torque that is produced.
Canadian Occupational Performance Measure | nine months
  Parents/caregivers and children choose 5 activities that they would like to see improve as a result of this intervention. The parent or caregiver rates how well their child currently performs that task and how satisfied they are with the performance of the task on a scale of 1-10 with 10 being the highest score.
Brain MRI - Diffusion tensor imaging | nine months
  A brain MRI scan is obtained. Tract based spatial statistics are performed from the scan to look for changes in individual voxels. Higher values for fractional anisotropy are associated with improved tract integrity. Lower values for radial and median diffusivity are associated with improved myelination.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen G Fowler, PhD, PT, Principal Investigator — University of California, Los Angeles
Locations (1):
- Center for Cerebral Palsy at UCLA/Orthopaedic Institute for Children, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vuong A, Joshi SH, Staudt LA, Matsumoto JH, Fowler EG. Improved Myelination following Camp Leg Power, a Selective Motor Control Intervention for Children with Spastic Bilateral Cerebral Palsy: A Diffusion Tensor MRI Study. AJNR Am J Neuroradiol. 2023 Jun;44(6):700-706. doi: 10.3174/ajnr.A7860. Epub 2023 May 4. PMID 37142433